CLINICAL TRIAL: NCT00599144
Title: Effectiveness for Postoperative Pain After Laparoscopic Cholecystectomy of 0,5% Bupivacaine-Soaked Tabotamp Placed in the Gallbladder Bed
Brief Title: Effectiveness of Bupivacaine After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Maria alla Gruccia Hospital (Other)
Responsible Party: Marco Scatizzi MD, Asl 8 santa maria alla gruccia hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: usl8
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Pain
Keywords: Cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Group1: a bupivacaine 0,5% (2mg/kg) soaked-tabotamp is placed in gallbladder bed after remove of gallbladder
  Interventions: Procedure: videolaparocholecystectomy
- 2 (Experimental): Group2: bupivacaine 0,5%(2mg/kg)is infiltrated in trocar incision after their closure.
  Interventions: Procedure: videolaparocholecystectomy
- 3 (No Intervention): Group3: control group without any local anesthetic use.
  Interventions: Procedure: videolaparocholecystectomy

INTERVENTIONS:
Procedure: videolaparocholecystectomy — Group1: a bupivacaine 0,5% (2mg/kg) soaked-tabotamp is placed in gallbladder bed after remove of gallbladder
  Arms: 1
Procedure: videolaparocholecystectomy — Group2: bupivacaine 0,5%(2mg/kg)is infiltrated in trocar incision after their closure.
  Arms: 1; 2
Procedure: videolaparocholecystectomy — Group3: control group without any local anesthetic use.
  Arms: 3

SUMMARY:
Evaluate the efficacy on postoperative pain of the positioning of a 0,5% bupivacaine soaked-tabotamp in gallbladder bed after videolaparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old, ASA 1 and 2
* Gallbladder adenomatous polyposis and cholelithiasis with no byochemical, clinical and instrumental evidence of acute cholecystitis at the moment of surgery.

Exclusion Criteria:

* Age<18 years old
* Pregnancy
* Previous major surgery of the supramesocholic compartment
* Acute cholecystitis
* Choledocolitiasis
* Acute pancreatitis at the moment of surgery
* Laparotomic conversion during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pain at 6 and 24 hours after surgery measured using the Visual Analogue Scale [VAS] [score 0 to 10, 0 = no pain, 10 = unbearable pain], | 6 and 24 hours after surgery

SECONDARY OUTCOMES:
Use of analgesics, extension of postsurgery hospitalization, post operative nausea and vomiting. | 6 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marco Scatizzi, MD, Principal Investigator — Ospedale Santa maria alla gruccia
Locations (1):
- Ospedale santa maria alla gruccia, Montevarchi, Ar, Italy

REFERENCES:
- [Background] Verma GR, Lyngdoh TS, Kaman L, Bala I. Placement of 0.5% bupivacaine-soaked Surgicel in the gallbladder bed is effective for pain after laparoscopic cholecystectomy. Surg Endosc. 2006 Oct;20(10):1560-4. doi: 10.1007/s00464-005-0284-5. Epub 2006 Aug 1. PMID 16897291
- [Derived] Feroci F, Kroning KC, Moraldi L, Borrelli A, Ottaviano A, De Prizio M, Scatizzi M. [A new effective method to reduce pain after laparoscopic cholecystectomy]. G Chir. 2010 Oct;31(10):423-8. Italian. PMID 20939947
- [Derived] Feroci F, Kroning KC, Scatizzi M. Effectiveness for pain after laparoscopic cholecystectomy of 0.5% bupivacaine-soaked Tabotamp placed in the gallbladder bed: a prospective, randomized, clinical trial. Surg Endosc. 2009 Oct;23(10):2214-20. doi: 10.1007/s00464-008-0301-6. Epub 2009 Jan 28. PMID 19184217